CLINICAL TRIAL: NCT04632849
Title: The Use of Libre to Educate, Motivate and Activate Adults With Newly Diagnosed Type 2 Diabetes to Improve Metabolic Control and Reduce Their Reliance on Medication: A Pilot Study
Brief Title: The Use of Libre to Improve Metabolic Control and Reduce Reliance on Medication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: University of Colorado, Denver (Other); West Virginia University (Other)
Responsible Party: Principal Investigator, Daniel Cox, PhD, Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22635
Record Dates: First submitted 2020-11-03; First posted 2020-11-17 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Intervention Model Description: All participants will receive the GEM intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GEM + CGM (Experimental): A self-directed lifestyle intervention for controlling Type 2 Diabetes
  Interventions: Behavioral: GEM + CGM

INTERVENTIONS:
Behavioral: GEM + CGM — Participants follow the GEM guidebook for 4 months (1 month of intervention and 3 months of maintenance) while wearing a FitBit activity monitor and a Freestyle Libre 2 CGM to provide feedback about activity and blood glucose. The GEM guidebook covers Routine choices, Recovering from blood glucose excursions, Reducing blood glucose excursions, and Maintenance.

SUMMARY:
GEM (Glycemic Excursion Minimization) is a new lifestyle treatment for type 2 diabetes that aims to lower glucose levels after meals and snacks. This is different from the current lifestyle treatment, which is to lose weight. This study is trying to find out if people who are newly diagnosed with type 2 diabetes can use a continuous glucose monitor together with the GEM lifestyle to improve control of their diabetes. Study participants will follow the GEM lifestyle for 4 months (1 month of treatment and 3 months of maintenance) instead of seeking usual care (medications or weight loss programs) to lower blood glucose.

DETAILED DESCRIPTION:
For people who are newly diagnosed with Type 2 Diabetes (T2D), it might be possible to delay or prevent the need for diabetic medications by reducing postprandial glucose (PPG). Our Glycemic Excursion Minimization (GEM) lifestyle intervention can reduce PPG, but it depends on blood glucose feedback to help the user learn what elevates their PPG. This study examines if continuous feedback from the Libre 2 continuous glucose monitor (CGM) will be advantageous for reaching the goals of GEM. We will recruit 18 adult participants newly diagnosed with type 2 diabetes who are interested in using the Libre 2 CGM. Six participants will be recruited from each of the primary care clinics at the University of Virginia (Dr. Cox), the University of Colorado (Dr. Oser) and the University of West Virginia, East Branch (Dr. Cucuzzella). Each site will also search their medical records to select 4 participants who match their study participants, meet the study criteria, but are being treated with routine care. These data will form the Routine Care control group (n=12). Routine Care participants will follow their doctor's treatment recommendations, while GEM participants will complete the 1-month, self-directed GEM lifestyle training using the Libre 2 CGM and a FitBit to monitor progress. They will then maintain the GEM lifestyle for 3 more months. The Total Treatment Effect (a measure of treatment effectiveness that considers both A1c and medication changes) will be calculated pre- and post-treatment from medical record data. CGM data from GEM participants will be collected and analyzed. CGM sensor use will be tracked to estimate participant engagement. We anticipate this multi-center pilot project will demonstrate the benefits of using Libre 2 with a structured lifestyle intervention designed to reduce postprandial blood glucose excursions for individuals newly diagnosed with T2D.

ELIGIBILITY:
Inclusion Criteria:(GEM group)

1. Provision of signed and dated informed consent form.
2. Willing to comply with study procedures and be available for the entire study.
3. 35 to 85 years of age, inclusive.
4. Diagnosed with Type 2 Diabetes within the last 12 months.
5. HbA1c between 6.5% and 11.5%.
6. Medical record contains HbA1c, lipid panel, BMI and blood pressure measures collected in the past three months.

Inclusion Criteria:(Routine Care group)

1. 35 to 85 years of age, inclusive.
2. Diagnosed with Type 2 Diabetes within the last 12 months.
3. HbA1c between 6.5% and 11.5%.
4. Medical record contains HbA1c, lipid panel, BMI and blood pressure measures collected in the past three months.

Exclusion Criteria (GEM group):

1. Has Type 1 Diabetes
2. Currently takes diabetes medication
3. Currently takes medication that can interfere with metabolic control, such as prednisone
4. Has a condition that precludes a low carbohydrate diet, such as gastroparesis
5. Has a physical or medical condition that precludes walking 120 steps per minute, for 10 minutes or longer
6. Has kidney disease.
7. Is receiving cancer treatment
8. Cannot speak English
9. Has blindness
10. Is pregnant or anticipates becoming pregnant in the next 4 months
11. Anticipates moving away within the next 4 months

Exclusion Criteria (Routine Care group): Individuals who met any of the following criteria in the first year after their T2D diagnosis will be excluded from the Routine Care group

1. Took medication that can interfere with metabolic control, such as prednisone
2. Had a condition that precludes a low carbohydrate diet, such as gastroparesis
3. Had a physical or medical condition that precludes walking 120 steps per minute, for 10 minutes or longer
4. Had kidney disease.
5. Was receiving cancer treatment
6. Was pregnant

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Total Treatment Effect (TTE) | Change from baseline TTE at 3 months post-intervention
  Measures the effect of the intervention on HbA1c. The TTE factors out the confounding effects of diabetes medications on HbA1c by adjusting for each medication's HbA1c-lowering equivalent.

SECONDARY OUTCOMES:
Blood glucose | Change from baseline blood glucose at 3 months post-intervention
  CGM measurement of blood glucose time in range, time above 150 mg/dL and time above 180 mg/dL Higher time in range means better outcomes.Higher time above 150 and 180 mg/dL means worse outcomes.
Physical activity | Change from baseline physical activity at 3 months post-intervention
  FitBit measurement of hours active, active minutes, and total steps. Higher activity means better outcomes.
Food Choice Questionnaire: High Glycemic Load (HGL) | Change from baseline Food Choice Questionnaire HGL at 3 months post-intervention
  Measures the servings of HGL foods eaten in a typical week. The scale ranges from 0 to no maximum. Higher scores mean worse outcomes.
Food Choice Questionnaire: Low Glycemic Load (LGL) | Change from baseline Food Choice Questionnaire LGL at 3 months post-intervention
  Measures the servings of LGL foods eaten in a typical week. The scale ranges from 0 to no maximum. Higher scores mean better outcomes.
Patient Health Questionnaire (PHQ-8) | Change from baseline PHQ-8 at 3 months post-intervention
  Measures depressive symptoms. The scale ranges from 0 to 24. Higher scores mean worse outcomes.
Diabetes Knowledge Scale | Change from baseline Diabetes Knowledge Scale at 3 months post-intervention
  Measures diabetes-related knowledge. The scale ranges from 0 to 26. Higher scores mean better outcomes.
Diabetes Empowerment Scale | Change from baseline Diabetes Empowerment Scale at 3 months post-intervention
  Measures the psychosocial self-efficacy of people with diabetes. The scale ranges from 0 to 40. Higher scores mean better outcomes.
Diabetes Distress Scale (Emotional Distress & Regimen Distress subscales) | Change from baseline Diabetes Distress Scale at 3 months post-intervention
  Measures concerns about diabetes. Each subscale ranges from 5 to 30. Higher scores mean worse outcomes.
Treatment Optimization Scale | Change from baseline Treatment Optimization Scale at 3 months post-intervention
  Generates user feedback about improving the intervention. The scale ranges from 43 to 215. Higher scores mean better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Cox, PhD, Principal Investigator — University of Virginia
Locations (1):
- Dept. of Psychiatry and Neurobehavioral Sciences, University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cox DJ, Banton T, Moncrief M, Conaway M, Diamond A, McCall AL. Minimizing Glucose Excursions (GEM) With Continuous Glucose Monitoring in Type 2 Diabetes: A Randomized Clinical Trial. J Endocr Soc. 2020 Aug 18;4(11):bvaa118. doi: 10.1210/jendso/bvaa118. eCollection 2020 Nov 1. PMID 33094208